CLINICAL TRIAL: NCT04276441
Title: HEARTLINE - A Heart Health Study Using Digital Technology to Investigate if Early AF Diagnosis Reduces the Risk of Thromboembolic Events Like Stroke IN the Real-world Environment
Brief Title: A Study to Investigate if Early Atrial Fibrillation (AF) Diagnosis Reduces Risk of Events Like Stroke in the Real-World
Status: Completed | Type: Observational
Sponsor: Janssen Scientific Affairs, LLC (Industry)
Collaborators: Apple Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108633; NOPRODAFL0002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2020-02-18; First posted 2020-02-19 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Non- Atrial Fibrillation (AF) Cohort: Participants without a history of AF will be randomly assigned into the study to either an Apple Watch/iPhone group or an iPhone group only.
  Interventions: Device: Heart healthy Engagement Program with the Apple Watch Series 5 or later
- Atrial Fibrillation (AF) Cohort: Participants with a diagnosis of AF taking a direct oral anti-coagulant (DOAC) for at least 30 days will be randomly assigned to Apple Watch/iPhone group or iPhone group only.
  Interventions: Device: Anti-Coagulation Adherence Module with the Apple Watch Series 5 or later

INTERVENTIONS:
Device: Heart healthy Engagement Program with the Apple Watch Series 5 or later — No drug will be given as part of this study. Participants without a diagnosis of AF will be enrolled and a heart healthy Engagement Program delivered via the Heartline app on the iPhone with the Apple Watch Series 5 or later.
  Groups: Non- Atrial Fibrillation (AF) Cohort
Device: Anti-Coagulation Adherence Module with the Apple Watch Series 5 or later — No drug will be given as part of this study. Participants with a diagnosis of AF (taking a DOAC for at least 30 days) will be enrolled and an Anti-Coagulation Adherence Module delivered via the Heartline app on the iPhone with an Apple Watch Series 5 or later.
  Groups: Atrial Fibrillation (AF) Cohort

SUMMARY:
The primary objectives of this study are to identify and diagnose Atrial Fibrillation (AF), evaluate improvement in cardiovascular (CV) outcomes, improve direct oral anti-coagulant (DOAC) adherence and persistence, and better characterize participants and identify predictors of disease.

ELIGIBILITY:
Inclusion Criteria:

* Medicare beneficiary either with Original or Medicare advantage
* Authorize electronic access to their healthcare claims data
* Authorize sharing of device sensor, health, and Heartline app data from their iPhone and Apple Watch (if applicable). This includes Apple Watch and iPhone sensor data that is not publicly available
* Willing and able to provide informed consent by electronically signing the remote e-consent directly in the Heartline app prior to any study-related activities. Electronically signing the remote e-consent indicates that he/she understands the purpose of, and activities required for the study and is willing to participate for the 2-year Active Engagement Phase, with continued passive collection of their device and healthcare claims data for an additional 1 year in the Post-Engagement Follow-Up Phase
* Current resident of the US at the time of eligibility screening, defined by self-reported state of residence within the 50 states or the US or District of Columbia
* Own an iPhone 6s or later with iOS Version 12.2 or later

Exclusion Criteria:

* Limited life expectancy and/or current diagnosis of terminal cancer
* Unable to confirm meeting inclusion criteria, including ability to consent and participate in human participant's research
* Own an Apple Watch Series 0 paired with an iPhone at the time of screening eligibility (these participants are not eligible for any study cohorts [randomized or observational])
* Have a confirmed diagnosis of Atrial Fibrillation (AF) at study entry and currently taking a direct oral anti-coagulant (DOAC) for less than (<) 30 days, currently taking other anti-coagulant medication(s) for AF other than a DOAC, or currently not taking medication for AF

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: The study population includes an older age group in whom the risk of developing Atrial Fibrillation (AF) is increased and who may benefit from a broad, health-focused Engagement Program paired with the irregular rhythm notification (IRN) alert (photoplethysmogram [PPG] sensor based) and electrocardiogram (ECG) sensor of the Apple Watch Series 5 or later.
Sampling Method: Probability Sample
Enrollment: 34244 (Actual)
Dates: Start 2020-02-25 (Actual); Primary Completion 2025-01-23 (Actual); Study Completion 2025-01-23 (Actual)

PRIMARY OUTCOMES:
Time from Randomization to Clinical Diagnosis of Atrial Fibrillation (AF) | Up to 3 years
  Time to a clinical diagnosis of AF obtained from healthcare claims database.
Percent Days Covered (PDC) by Direct Oral Anti-Coagulant (DOAC) Prescription Fills | Up to 3 years
  Percent days of covered prescription DOAC use minus any evidence of no prescription use/refills over the time interval chosen.

SECONDARY OUTCOMES:
Time to Composite of 6-component Events (Ischemic Stroke/TIA, MI, Non-CNS Embolism or Thrombosis, Hospitalization or ED Visit for HF, CV Hospitalization and ACM) | Up to 3 years
  Time to composite of 6-component events (ischemic stroke/transient ischemic attack [TIA], myocardial infarction [MI], non-central nervous system [CNS] embolism or thrombosis, hospitalization or emergency department [ED] visit due to heart failure [HF], cardiovascular [CV] hospitalization, and all-cause mortality [ACM]), obtained from randomization in the healthcare claims database, will be reported.
Summary of Total Cost of Care Delivery, Total Health Resource Utilization (HRU), and Cost Effectiveness | Up to 3 years
  Summary of total cost of care delivery, total HRU, and cost effectiveness will be reported. Total costs of care reported as number of HRU events times the unit cost for each event. HRU reported as counts of HRU events. Cost effectiveness to be assessed by including the cost to diagnosis, treatment and reported clinical outcome.
Time to Ischemic stroke/TIA | Up to 3 years
  Ischemic stroke/TIA is defined as a hospitalization/diagnosis for Ischemic stroke/TIA.
Time to MI | Up to 3 years
  MI is defined as a hospitalization/diagnosis for MI.
Time to non-CNS Embolism or Thrombosis | Up to 3 years
  Non-CNS embolism or thrombosis is defined as hospitalization for non-CNS thromboembolic events.
Time to Hospitalization or ED for HF | Up to 3 years
  Hospitalization or ED visit for HF is defined as an in-patient stay or an outpatient ED visit for HF.
Time to CV Hospitalization | Up to 3 years
  Hospitalization for CV is defined as an in-patient stay for CV disease.
Time to all-Cause Mortality | Up to 3 years
  All-cause mortality (ACM) is defined as deaths from all (reported) causes.
Time to Composite Bleeding Events Resulting in Hospitalization | Up to 3 years
  Hospitalization for composite bleeding events (such as intracranial hemorrhage, gastrointestinal [GI], respiratory, intraocular) is defined as in-patient stay for bleeding events, as reported in the healthcare claims database.
Time to Hospitalization for Hemorrhagic Stroke | Up to 3 years
  Hospitalization for hemorrhagic stroke is defined as an in-patient stay for a hemorrhagic stroke.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Scientific Affairs, LLC Clinical Trial, Study Director — Janssen Scientific Affairs, LLC
Locations (1):
- Evidation Health, San Mateo, California, United States

REFERENCES:
- [Derived] Nikolovski J, Navar AM, Steinhubl S, Baca-Motes K, Curtis AB, Peterson ED, Lakkireddy D, Tarino M, Juan S, Damaraju CRV, Wentworth D, Wildenhaus K, Patel M, Tavakoli C, Gibson CM, Spertus JA; Heartline Steering Committee. The Heartline Experience: Achieving Long-Term Participant Engagement in Digital Health Technology Trials. JACC Adv. 2025 Sep;4(9):102072. doi: 10.1016/j.jacadv.2025.102072. Epub 2025 Aug 20. PMID 40839901
- [Derived] Gibson CM, Steinhubl S, Lakkireddy D, Turakhia MP, Passman R, Jones WS, Bunch TJ, Curtis AB, Peterson ED, Ruskin J, Saxon L, Tarino M, Tarakji KG, Marrouche N, Patel M, Harxhi A, Kaul S, Nikolovski J, Juan S, Wildenhaus K, Damaraju CV, Spertus JA; Heartline Steering Committee. Does early detection of atrial fibrillation reduce the risk of thromboembolic events? Rationale and design of the Heartline study. Am Heart J. 2023 May;259:30-41. doi: 10.1016/j.ahj.2023.01.004. Epub 2023 Jan 12. PMID 36642226
- [Derived] Nikolovski J, Koldijk M, Weverling GJ, Spertus J, Turakhia M, Saxon L, Gibson M, Whang J, Sarich T, Zambon R, Ezeanochie N, Turgiss J, Jones R, Stoddard J, Burton P, Navar AM. Factors indicating intention to vaccinate with a COVID-19 vaccine among older U.S. adults. PLoS One. 2021 May 24;16(5):e0251963. doi: 10.1371/journal.pone.0251963. eCollection 2021. PMID 34029345